CLINICAL TRIAL: NCT00926783
Title: Selective CFAE Targeting for Atrial Fibrillation (SELECT-AF)
Brief Title: Selective Complex Fractionated Atrial Electrograms (CFAE) Targeting for Atrial Fibrillation
Acronym: SELECT-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SELECT-AF
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Atrial Fibrillation
Keywords: paroxysmal; persistent; targeted; generalized; CFAE
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- (1) targeted CFAE ablation (Active Comparator)
  Interventions: Procedure: CFAE ablation
- (2) generalized CFAE ablation (Active Comparator)
  Interventions: Procedure: CFAE ablation

INTERVENTIONS:
Procedure: CFAE ablation — CFAE ablation (targeted vs. generalized)
  Other Names: CFAE ablation (targeted vs. generalized); NaviStar ThermoCool Catheter; CARTO mapping system

SUMMARY:
This study will be a multicenter, open, prospective, randomized trial. Patients with either paroxysmal or persistent atrial fibrillation will be considered for the study. (For US, only paroxysmal atrial fibrillation will be considered.) Eligible subjects will be randomized into one of two arms in the study: (1) targeted CFAE ablation or (2) generalized CFAE ablation. Both techniques will then be followed by PVAI (pulmonary vein antral isolation) as part of a hybrid ablation strategy. The nature of the ablation procedures does not allow physicians to be blinded to the randomization.

DETAILED DESCRIPTION:
The purpose of this study is to compare a strategy of targeted CFAE ablation, focusing on regions of continuous electrical activity versus a strategy of generalized CFAE ablation in terms of (1) acute effects on AFCL (atrial fibrillation cycle length), AF regularization, and AF termination; (2) number and distribution of lesion sets delivered; and (3) long term effects on procedural outcome when combined with PVAI as a hybrid strategy.

ELIGIBILITY:
Inclusion Criteria:

Candidates for this study must meet ALL of the following criteria:

* Age ≥ 18 years old
* First-time ablation procedure for AF
* Symptomatic AF which has been refractory to at least one antiarrhythmic medication (AAD). "Symptomatic" patients are those who have been aware of their AF anytime within the last 5 years. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, or other symptoms, or any combination of the above
* One of the following must apply:

  * AF must either be PERSISTENT AF (non-US sites only) or HIGH BURDEN PAROXYSMAL AF - High burden paroxysmal AF is defined as episodes that terminate within 30 days and meet any ONE of the following criteria:
  * More than 1 episode of AF per month in the preceding 6 months with at least 1 episode lasting >24 hours by symptoms,
  * LA size of >/= 48 mm in the PLAX (parasternal long axis) view on echocardiography
  * LA volume >/= 100 cc
  * Total AF history >/= 10 years
* At least one episode of AF must have been documented by ECG, Holter, TTM, or telemetry strip within 24 months of inclusion in the study.
* Patients must be able and willing to provide written informed consent to participate in the study.
* Able and willing to comply with all pre-, post- and follow-up testing and requirements.

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions apply:

* Patients with long-standing persistent AF >1 year for which cardioversion (pharmacologic or electrical) has failed or will never be attempted.
* Patients with AF felt to be secondary to an obvious reversible cause.
* Patients with contraindications to systemic anticoagulation with heparin or Coumadin.
* Patients who have previously undergone atrial fibrillation ablation.
* Patients who are pregnant (by history of menses or pregnancy test if history is considered unreliable.
* Left atrial size ≥55 mm (PLAX view on echocardiography).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-08; Primary Completion 2011-11 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hendricks, Study Director — Biosense Webster, Inc.
Locations (7):
- United States (2):
  - Loyola University Medical Center, Maywood, Illinois
  - Johns Hopkins University, Baltimore, Maryland
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Canada (4):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Southlake Regional Health Center, Newmarket, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital Laval - Institut universitaire de cardiologie et de pneumonologie, Québec, Quebec

REFERENCES:
- [Derived] Verma A, Sanders P, Champagne J, Macle L, Nair GM, Calkins H, Wilber DJ. Selective complex fractionated atrial electrograms targeting for atrial fibrillation study (SELECT AF): a multicenter, randomized trial. Circ Arrhythm Electrophysiol. 2014 Feb;7(1):55-62. doi: 10.1161/CIRCEP.113.000890. Epub 2014 Jan 14. PMID 24425420

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject of the study was consented on August 17, 2009. The final follow-up was performed on November 14, 2011. The total study duration was approximately 27 months. A total of 86 subjects were enrolled from 7 participating sites; 2 sites in the United States (US), 4 sites in Canada, and 1 site in Australia.
Pre-assignment Details: Among the 86 consented subjects, two were excluded prior to randomization; one was excluded due to thrombus found on pre-procedure echo. Hence only 83 subjects were randomized to the two treatment arms and underwent radio-frequency ablation
Groups:
- Targeted CFAE Ablation: Targeted complex fractionated atrial electrograms (CFAE) ablation focuses on highly selective regions of continuous electrical activity (CEA) that are critical to Atrial Fibrillation (AF) perpetuation. In the Targeted arm, the cardiac mapping system collects the abnormal electrical heart signals that are displayed in another specific color when the abnormal electrical signal is above the normal for more than the specified percentage of time over a pre-specified length of time.
- Generalized CFAE Ablation: Generalized complex fractionated atrial electrograms (CFAE) ablation focused on all repetitive CAFE, which was defined as interval confidence level (ICL) > 5. In the Generalized arm, the cardiac mapping system collects the abnormal electrical heart signals and displays in a specific color when the number of electrical signals are more than the specified number over a pre-specified length of time.
Period: Overall Study
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Started | 42 | 41
Completed | 39 | 38
Not Completed | 3 | 3
Not completed — Incomplete CFAE Procedures | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is based on enrolled subjects (86) who had demographic information. Four subjects, who didn't have demographic data, were excluded from baseline analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.8) | 61.5 (9.2) | 61.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 29 | 31 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 37 | 32 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 12
Atrial fibrillation type [Number; unit: participants]
  High Burden Paroxysmal | 11 | 19 | 30
  Persistent | 31 | 21 | 52
Duration of Atrial fibrillation diagnosis (Year) [Mean (Standard Deviation); unit: years] | 5.8 (5.7) | 5.2 (5.2) | 5.5 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Were Free From Atrial Arrhythmia at One Year.
Description: Proportion of subjects who were free from atrial arrhythmia (no recurrence of atrial fibrillation, atrial flutter, and atrial tachycardia (AF/AFL/AT)) between Day 91 and Day 365 post first ablation procedure.
Time Frame: From day 91 to day 365 post first ablation procedure
Population: Per-protocol population - subjects who underwent repeat ablation procedures within six months of initial procedures.
Measure: Number; unit: participants
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Number analyzed (Participants) | 39 | 38
participants
  Without recurrence AF/AFL/AT | 10 | 18
  With recurrence AF/AFL/AT | 29 | 20
Statistical Analysis 1: Comparison: Targeted CFAE Ablation vs Generalized CFAE Ablation; The null hypothesis is that rates of free from atrial arrhythmia for the two arms, Targeted and Generalized, are the same. The alternative hypothesis is that the rates are not the same. Due to the lack of literature data comparing these endpoints between two randomization groups, the sample size is not statistically powered to support statistical inferences; Test type: Superiority or Other; p = 0.048, Fisher Exact — The p-value was based on Fisher's exact test. There were no adjustments for multiple comparisons

2. Primary Outcome: Total Radio-frequency (RF) Delivery Time During CFAE
Description: Total RF delivery time (minutes) is defined as the duration of the RF delivered per ablation site and totaled for each procedure.
Time Frame: Duration of an Atrial Fibrillation RF ablation procedure (up to about 5 hours)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Number analyzed (Participants) | 39 | 37
Minutes | 23.2 (19.7) | 37.8 (20.1)
Statistical Analysis 1: Comparison: Targeted CFAE Ablation vs Generalized CFAE Ablation; The null hypothesis is that the total RF delivery times for both arms are equal. The alternative hypothesis is that the total RF delivery times are not equal. Due to the lack of literature data comparing these endpoints between two randomization groups, the sample size is not statistically powered to support statistical inferences; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

3. Secondary Outcome: Duration of Ablation Procedure
Description: Duration of ablation procedure includes three components: Access time - Time from first stick to tracking of the NAVISTAR catheter to the chamber of interest; Mapping time - Creation of first workable map; Ablation and verification time - Creation and verification of all ablation points including pulmonary vein isolation and complex fractionated electrograms.
Time Frame: Duration of ablation procedure (up to about 5 hours)
Population: Per-protocol population with available outcome data
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Number analyzed (Participants) | 39 | 38
Minutes
  Total Procedure Time | 220.6 (59.4) | 226.1 (52.0)
  Procedure Time to Access Site | 42.7 (20.8) | 45.4 (22.4)
  Procedure Time to Mapping | 35.7 (26.5) | 27.4 (10.5)
  Procedure Time to Ablation and Verification | 132.8 (43.0) | 149.9 (47.7)

4. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy time is divided into: Fluoroscopy time for access - Time to track the NAVISTAR catheter to the chamber of interest; Fluoroscopy time to map - Creation of first workable map, ablation, and verification time; Fluoroscopy to create and verify all ablation points including pulmonary vein isolation and complex fractionated electrograms.
  Fluoroscopy time for access is independent of the strategies and will not be included in comparative analysis.
Time Frame: Duration of an Atrial Fibrillation RF ablation procedure (up to about 5 hours)
Population: Per-protocol population with available outcome data
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Number analyzed (Participants) | 39 | 38
Minutes
  Total Fluoroscopy Time | 57.4 (20.2) | 60.1 (19.3)
  Fluoroscopy Time to Gain Access | 9.7 (8.3) | 11.8 (11.6)
  Fluoroscopy Time to Mapping | 15.5 (12.6) | 13.8 (11.1)
  Fluoroscopy Time to Ablation and Verification | 36.9 (10.9) | 41.5 (22.1)

5. Secondary Outcome: Change in Atrial Fibrillation Cycle Length From Baseline to the End of the Ablation Procedure for Each Target
Description: Change in atrial fibrillation cycle length from baseline to the end of the ablation procedure for each target
Time Frame: Duration of an Atrial Fibrillation RF ablation procedure (up to 5 hours)
Population: Per-protocol population with available outcome data
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Number analyzed (Participants) | 38 | 38
Milliseconds | 23.3 (33.3) | 25.4 (32.8)

6. Secondary Outcome: Incidence of Atrial Fibrillation (AF) Termination/Regularization
Description: Incidence of Atrial Fibrillation (AF) termination/regularization is defined as AF terminates during a complex fractionated atrial electrograms (CFAE) procedure.
Time Frame: Duration of an Atrial Fibrillation RF ablation procedure (up to about 5 hours)
Population: Per-protocol population with available outcome data
Measure: Number; unit: participants
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Number analyzed (Participants) | 39 | 38
participants | 11 | 14

ADVERSE EVENTS:
Time Frame: 12 months post procedure follow up.
Arm/Group | Targeted CFAE Ablation | Generalized CFAE Ablation
Serious Adverse Events (participants affected / at risk) | 15/42 | 11/41
Other Adverse Events (participants affected / at risk) | 29/42 | 31/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted CFAE Ablation (N=42) | Generalized CFAE Ablation (N=41)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (2)
Atrial Flutter (Cardiac disorders) | 2 (5) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Heart Block (Cardiac disorders) | 0 (0) | 1 (1)
Pacemaker (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Node Disease (Cardiac disorders) | 2 (2) | 0 (0)
Sinus Node Injury (Cardiac disorders) | 1 (1) | 0 (0)
Tachy-Brady Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (General disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Pruritus (General disorders) | 1 (1) | 0 (0)
Parasite (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vocal Chord Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Targeted CFAE Ablation (N=42) | Generalized CFAE Ablation (N=41)
Angina Pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (5) | 8 (9)
Atrial Flutter (Cardiac disorders) | 6 (6) | 7 (7)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardioversion (Cardiac disorders) | 2 (2) | 0 (0)
Chest Discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Medication Reaction (Cardiac disorders) | 1 (2) | 0 (0)
Mild Blunting (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 4 (4) | 3 (3)
Pericardial Separation (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (3)
Tachycardia NEC (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract Surgery (Eye disorders) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 1 (1)
Visual Disturbance or Impairment (Eye disorders) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatitis (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fluid Overload (General disorders) | 0 (0) | 1 (1)
Hematoma (General disorders) | 3 (5) | 3 (3)
Localized Edema (General disorders) | 1 (1) | 0 (0)
Low Potassium (General disorders) | 1 (1) | 0 (0)
Medication Reaction (General disorders) | 1 (1) | 0 (0)
Pedial Edema (General disorders) | 1 (1) | 0 (0)
Post Procedural Elevated Blood Sugar (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 1 (1)
Rash (General disorders) | 1 (1) | 0 (0)
Wound Complication (General disorders) | 1 (1) | 0 (0)
Elevated Liver Enzymes (Hepatobiliary disorders) | 0 (0) | 1 (1)
Shingles (Immune system disorders) | 1 (1) | 0 (0)
Dysuria (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Anesthesia Complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Glossodynia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Groin Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 8 (8)
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Ruptured Tendon (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 2 (2) | 3 (3)
Trouble Concentrating (Nervous system disorders) | 1 (1) | 0 (0)
Vasovagal Response (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Increased Urine Output (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Phrenic Nerve Damage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is allowed to publish but must submit draft pubs to Biosense Webster, Inc. at least 30 days prior to submission for publication or presentation.